CLINICAL TRIAL: NCT04939285
Title: Effect of PEEP=5cmH2O vs PEEP=0cmH2O PSV Strategies During SBT on Successful Disconnection From Mechanical Ventilation: A Randomized Clinical Trial
Brief Title: Effect of PEEP=5cmH2O vs PEEP=0cmH2O PSV Strategies During SBT on Successful Disconnection From Mechanical Ventilation
Acronym: PPSDMV-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu ZiMeng, associate professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020761001
Record Dates: First submitted 2020-06-07; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Respiration, Artificial
Keywords: PEEP; pressure support ventilation; SBT
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP=5cmH2O (Experimental): In PSV mode,PS = 8 cmH2O,PEEP= 5 cmH2O, and FiO2 level was consistent with that before SBT
  Interventions: Procedure: PEEP
- PEEP=0cmH2O (Experimental): In PSV mode,PS = 8 cmH2O,PEEP=0 cmH2O, and FiO2 level was consistent with that before SBT
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: PEEP — The patients who met the withdrawal screening criteria were randomly divided into low pressure support level PSV spontaneous respiration test.The duration of the spontaneous breathing test was 30 minutes, and the results of the spontaneous breathing test were evaluated at the end of the test.

SUMMARY:
Mechanical ventilation is the most common means of life support in intensive care unit. Daily spontaneous breathing trial (SBT) is the most effective method to evaluate whether patients on mechanical ventilation can be removed from the ventilator, thus reducing mechanical ventilation duration and ventilator-related complications. Pressure support ventilation and T-piece ventilation are the two most commonly used SBT methods, lasting from 30 minutes to 2 hours. However, the parameter setting for SBT using PSV method has not been completely agreed, especially regarding the use of positive end-expiratory pressure (PEEP). Therefore, we intend to conduct a single-center, prospective, randomized, controlled study to evaluate the impact of PEEP=0cmH2O and PEEP=5cmH2O on extubation success rate and re-intubation rate in mechanically ventilated patients, to provide high-level clinical evidence on the use of PEEP for SBT in patients with mechanical ventilation, so as to reduce the duration of mechanical ventilation and complications related to mechanical ventilation.

DETAILED DESCRIPTION:
Patients who met the withdrawal screening criteria were randomly divided into groups for self-breathing test by PSV method with low pressure support level. Parameters of each group were as follows. In the experimental group, PS = 8 cmH2O, PEEP= 5 cmH2O, and FiO2 level was consistent with that before SBT.The control group: PSV mode, PS = 8 cmH2O, PEEP=0 cmH2O, FiO2 level was consistent with that before SBT.The duration of the spontaneous breathing test was 30 minutes, and the results of the spontaneous breathing test were evaluated at the end of the test.Endotracheal intubation was removed if the patient was successfully assessed for spontaneous breathing. Record the date and time of extubation.Patients with endotracheal intubation were treated with nasal hyperflow oxygen therapy for respiratory support.Patients with SBT failure were reconnected to the ventilator, and mechanical ventilation was given according to the ventilation mode and parameters before the spontaneous breathing test.The reasons for SBT failure were recorded and these patients were not randomized to SBT.If respiratory failure occurs within 48 hours after extubation, the attending physician decides the respiratory treatment plan.These patients were also not included in the subsequent SBT randomization.

ELIGIBILITY:
Inclusion Criteria:

* 1) Older than 18;
* 2) Patients with mechanical ventilation for 24h;
* 3) Meet the screening standards for daily disconnection;
* 4) The study complies with the Declaration of Helsinki and China's regulations on clinical trial research, and the patient or his/her family members have informed and agreed to participate in the study.

Exclusion Criteria:

* 1) Patients undergoing tracheotomy;
* 2) Patients who refuse to be intubated again after endotracheal intubation is removed;
* 3) Patients on long-term mechanical ventilation: mechanical ventilation duration was continuous for 21 days, >6 h/d;
* 4) The attending physician decides the withdrawal plan (e.g., the potential pathology is more favorable to the specific withdrawal plan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Extubation success rate | during 48 hours after the first SBT
  The success rate of extubation (during 48 hours after the first SBT if successfully removed from the ventilator).
Reintubation rate | during 48 hours after extubation
  The reintubation rate of respiratory failure after extubation.

SECONDARY OUTCOMES:
Reintubation rate at 72 hours | during 72 hours after extubation
  Reintubation rate at 72 h
No mechanical ventilation duration in ICU | From first transfer in ICU to transfer out ICU up to 28 days after randomization
  No mechanical ventilation duration in ICU
Length of ICU stay | From admission to discharge from ICU up to 28 days after randomization
  Length of ICU stay
ICU mortality, 28-day mortality | 28 day
  ICU mortality, 28-day mortality
Results of blood gas analysis | every 30 min during SBT up one hour to and 30min after extubation
  PaCO2 and PaO2 (SBT screening, SBT completion, 30min after extubation)
Respiratory mechanical parameters | every 30 min during SBT up to one hour
  lung compliance monitoring： Static and dynamic lung compliance
Predictors of withdrawal of patients on mechanical ventilation | every 30 min during SBT up one hour and before extubation
  airway occlusion pressure
Predictors of withdrawal of patients on mechanical ventilation | every 30 min during SBT up one hour and before extubation
  negativeinspiratory force
Predictors of withdrawal of patients on mechanical ventilation | every 30 min during SBT up to one hour and before extubation
  Rapid Shallow Breathing Index
Vital signs | every 15 min during SBT up to one hour and 30 min after extubation
  Heart Rate
Vital signs | every 15 min during SBT up to one hour and 30 min after extubation
  SpO2
Vital signs | every 15 min during SBT up to one hour and 30 min after extubation
  Blood Pressure

OTHER OUTCOMES:
Chest electrical impedance imaging (EIT) | from the start to the end of SBT up to one hour and 30min after extubation
  region of interests(RI),Center of Ventilation(COV),end expiratory lung inmpedance(EELI), △EELi
Subjective score of patients with dyspnea | every 30 min during SBT up to one hour and 30min after extubation
  Score 0-10: 0 for no dyspnea, 10 for severe dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: ZiMeng Liu, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The first affiliated hospital of SunYatSen University, Guanzhou, Guangdong, China

REFERENCES:
- [Background] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Background] Esteban A, Alia I, Tobin MJ, Gil A, Gordo F, Vallverdu I, Blanch L, Bonet A, Vazquez A, de Pablo R, Torres A, de La Cal MA, Macias S. Effect of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation. Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1999 Feb;159(2):512-8. doi: 10.1164/ajrccm.159.2.9803106. PMID 9927366
- [Background] Perren A, Domenighetti G, Mauri S, Genini F, Vizzardi N. Protocol-directed weaning from mechanical ventilation: clinical outcome in patients randomized for a 30-min or 120-min trial with pressure support ventilation. Intensive Care Med. 2002 Aug;28(8):1058-63. doi: 10.1007/s00134-002-1353-z. Epub 2002 Jul 13. PMID 12185425
- [Background] Sklar MC, Burns K, Rittayamai N, Lanys A, Rauseo M, Chen L, Dres M, Chen GQ, Goligher EC, Adhikari NKJ, Brochard L, Friedrich JO. Effort to Breathe with Various Spontaneous Breathing Trial Techniques. A Physiologic Meta-analysis. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1477-1485. doi: 10.1164/rccm.201607-1338OC. PMID 27768396
- [Background] Pellegrini JA, Moraes RB, Maccari JG, de Oliveira RP, Savi A, Ribeiro RA, Burns KE, Teixeira C. Spontaneous Breathing Trials With T-Piece or Pressure Support Ventilation. Respir Care. 2016 Dec;61(12):1693-1703. doi: 10.4187/respcare.04816. Epub 2016 Sep 6. PMID 27601720
- [Background] Burns KEA, Soliman I, Adhikari NKJ, Zwein A, Wong JTY, Gomez-Builes C, Pellegrini JA, Chen L, Rittayamai N, Sklar M, Brochard LJ, Friedrich JO. Trials directly comparing alternative spontaneous breathing trial techniques: a systematic review and meta-analysis. Crit Care. 2017 Jun 1;21(1):127. doi: 10.1186/s13054-017-1698-x. PMID 28576127
- [Background] Li Y, Li H, Zhang D. Comparison of T-piece and pressure support ventilation as spontaneous breathing trials in critically ill patients: a systematic review and meta-analysis. Crit Care. 2020 Feb 26;24(1):67. doi: 10.1186/s13054-020-2764-3. PMID 32102693
- [Background] Subira C, Hernandez G, Vazquez A, Rodriguez-Garcia R, Gonzalez-Castro A, Garcia C, Rubio O, Ventura L, Lopez A, de la Torre MC, Keough E, Arauzo V, Hermosa C, Sanchez C, Tizon A, Tenza E, Laborda C, Cabanes S, Lacueva V, Del Mar Fernandez M, Arnau A, Fernandez R. Effect of Pressure Support vs T-Piece Ventilation Strategies During Spontaneous Breathing Trials on Successful Extubation Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jun 11;321(22):2175-2182. doi: 10.1001/jama.2019.7234. PMID 31184740
- [Background] Schmidt GA, Girard TD, Kress JP, Morris PE, Ouellette DR, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Truwit JD. Liberation From Mechanical Ventilation in Critically Ill Adults: Executive Summary of an Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline. Chest. 2017 Jan;151(1):160-165. doi: 10.1016/j.chest.2016.10.037. Epub 2016 Nov 3. PMID 27818329
- [Background] El-Khatib MF, Zeineldine SM, Jamaleddine GW. Effect of pressure support ventilation and positive end expiratory pressure on the rapid shallow breathing index in intensive care unit patients. Intensive Care Med. 2008 Mar;34(3):505-10. doi: 10.1007/s00134-007-0939-x. Epub 2007 Dec 1. PMID 18060662
- [Background] Futier E, Constantin JM, Petit A, Jung B, Kwiatkowski F, Duclos M, Jaber S, Bazin JE. Positive end-expiratory pressure improves end-expiratory lung volume but not oxygenation after induction of anaesthesia. Eur J Anaesthesiol. 2010 Jun;27(6):508-13. doi: 10.1097/EJA.0b013e3283398806. PMID 20404729
- [Background] Ostberg E, Thorisson A, Enlund M, Zetterstrom H, Hedenstierna G, Edmark L. Positive End-expiratory Pressure Alone Minimizes Atelectasis Formation in Nonabdominal Surgery: A Randomized Controlled Trial. Anesthesiology. 2018 Jun;128(6):1117-1124. doi: 10.1097/ALN.0000000000002134. PMID 29462011
- [Background] Young CC, Harris EM, Vacchiano C, Bodnar S, Bukowy B, Elliott RRD, Migliarese J, Ragains C, Trethewey B, Woodward A, Gama de Abreu M, Girard M, Futier E, Mulier JP, Pelosi P, Sprung J. Lung-protective ventilation for the surgical patient: international expert panel-based consensus recommendations. Br J Anaesth. 2019 Dec;123(6):898-913. doi: 10.1016/j.bja.2019.08.017. Epub 2019 Oct 3. PMID 31587835
- [Background] Cabello B, Thille AW, Roche-Campo F, Brochard L, Gomez FJ, Mancebo J. Physiological comparison of three spontaneous breathing trials in difficult-to-wean patients. Intensive Care Med. 2010 Jul;36(7):1171-9. doi: 10.1007/s00134-010-1870-0. Epub 2010 Mar 30. PMID 20352189
- See also: Related Info — http://www.nejm.org/doi/full/10.1056/NEJM199502093320601
- See also: Related Info — http://www.nejm.org/doi/full/10.1056/NEJM199612193352502
- See also: Related Info — http://www.atsjournals.org/doi/full/10.1164/ajrccm.159.2.9803106
- See also: Related Info — http://link.springer.com/article/10.1007%2Fs00134-002-1353-z
- See also: Related Info — http://ccforum.biomedcentral.com/articles/10.1186/s13054-017-1698-x
- See also: Related Info — http://ccforum.biomedcentral.com/articles/10.1186/s13054-020-2764-3
- See also: Related Info — http://jamanetwork.com/journals/jama/fullarticle/2735502
- See also: Related Info — http://linkinghub.elsevier.com/retrieve/pii/S0012369216623255
- See also: Related Info — http://link.springer.com/article/10.1007%2Fs00134-007-0939-x
- See also: Related Info — http://journals.lww.com/ejanaesthesiology/toc/9000/00000
- See also: Related Info — http://journals.lww.com/pages/default.aspx
- See also: Related Info — http://link.springer.com/article/10.1007%2Fs00134-010-1870-0